CLINICAL TRIAL: NCT03898908
Title: Phase II, Multicentre Clinical Trial to Evaluate the Activity of Encorafenib and Binimetinib Administered Before Local Treatment in Patients With BRAF Mutant Melanoma Metastatic to the Brain
Brief Title: Encorafenib and Binimetinib Before Local Treatment in Patients With BRAF Mutant Melanoma Metastatic to the Brain
Acronym: EBRAIN-MEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: Pierre Fabre Medicament (Industry); MFAR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-1802; 2018-002530-20 (EudraCT Number)
Record Dates: First submitted 2019-03-27; First posted 2019-04-02 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Melanoma; Brain Metastases
Keywords: metastases; melanoma; encorafenib; binimetinib
MeSH Terms: conditions — Melanoma; Brain Neoplasms; Neoplasm Metastasis | interventions — encorafenib; binimetinib; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Cohort 1 will include patients with asymptomatic brain metastases and without previous local treatment in the brain (N=48), while cohort 2 will include patients with symptomatic brain metastasis and without previous local treatment in the brain (N=15).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COMBO450 (Experimental): Encorafenib - Orally, 75 mg and 50 mg capsules Binimetinib - Orally, 15 mg tablets
  In each cohort, patients will be treated with encorafenib 450 mg once daily and binimetinib 45 mg twice daily until PD or death.
  Interventions: Drug: encorafenib; Drug: binimetinib; Radiation: Whole brain radiation therapy; Radiation: Radiosurgery/stereotactic radiosurgery

INTERVENTIONS:
Drug: encorafenib — Encorafenib 75mg and 50mg (capsules) for a 450mg daily for oral administration during 56 days and after local radiation treatment.
  If no progression of disease progression (PD) is reported, treatment will continue until PD, unacceptable toxicity or death.
  Other Names: Braftovi
Drug: binimetinib — Binimetinib 15mg (tablets) for a 45mg/12 hours for oral administration during 56 days and after local radiation treatment.
  Other Names: Mektovi
Radiation: Whole brain radiation therapy — The whole brain planning target volume (PTV) will receive 30 Gy in 10 fractions.
  Treatment will be delivered once daily, 5 fractions per week, over 2 to 2.5 weeks.
Radiation: Radiosurgery/stereotactic radiosurgery — Dose selection must be based on previously published Radiation Therapy Oncology Group (RTOG) data, with dose modification left up to the treating physician. The total dose will depend on the size of the metastatic lesion(s) and proximity to critical structures.
  Suggested doses are as follow: 1 fraction x 15-25 Gy; 3 fractions x 9-11 Gy; 5 fractions x 6-7 Gy; or 6 fractions x 5-6 Gy.
  For GTV > 20 mm hypofractionated stereotactic radiotherapy could be preferred. Treatment will be delivered once daily, alternate-day, 3 fractions per week.

SUMMARY:
Phase II clinical trial, with two cohorts of patients included in parallel, all with melanoma BRAF mutated and brain metastases without previous local treatment in the brain. Cohort 1 will include patients with asymptomatic brain metastases and cohort 2 will include patients with symptomatic brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of approved by the investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to the performance of any trial activities.
* Histologically confirmed diagnosis of unresectable metastatic cutaneous melanoma, or unknown primary melanoma with one or more brain metastasis with a diameter of 10 to 50 mm, measured by contrast enhanced MRI.
* Presence of a BRAF V600E or V600K mutation, or both, in their tumour tissue.
* Barthel Index of Activities of Daily Living > 10.
* Subjects aged ≥ 18 years.
* ECOG 0-1 in asymptomatic patients (cohort 1), 0-2 in symptomatic patients (cohort 2).
* Adequate haematological function (Haemoglobin ≥ 9 g/dL, may have been transfused; Platelet count ≥ 100 × 109/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.)
* Adequate hepatic function defined by a total bilirubin level ≤ 2.0 × the upper limit of normality (ULN) and AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
* Serum Creatinine ≤ 2.0 x ULN or estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
* Evidence of at least one measurable lesion as detected by radiological or photographic methods according to guidelines based on Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
* Naïve untreated patients or patients who have progressed on or after prior first line immunotherapy for unresectable locally advanced or metastatic melanoma, but it must have ended at least 6 weeks prior to randomization; prior adjuvant therapy is permitted (e.g. IFN, IL-2 therapy, any other immunotherapy, radiotherapy or chemotherapy), BRAF or MEK inhibitors can be used in the adjuvant setting, providing the relapse does not occur during the adjuvant treatment or within 12 months after the end of it, and providing the adjuvant treatment with targeted therapy did not cause in the patient any grade 3-4 toxicity not including medically serious and reversible/controlled toxicities (ex: GGT elevation, CPK elevation, vomiting).
* Steroids or anticonvulsants are allowed if clinically needed and are not being administered in an increasing dose.
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Normal functioning of daily living activities.
* Willingness and ability to attend scheduled visits, follow the treatment schedule and undergo clinical tests and other study procedures.

Exclusion Criteria:

* Uveal or mucosal melanoma.
* History of leptomeningeal metastases, with the exception that they are only seen in brain MRI and the patient has ECOG 0-1 and no neurological symptoms (except for cohort 2, where symptomatic patients will be allowed if ECOG is 0-2).
* Another cancer in the last five years, except for in situ carcinoma of the cervix or squamous cell carcinoma of the skin adequately treated or limited basal cell skin cancer adequately controlled.
* History of or current evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO) or history of retinal degenerative disease (RDD).
* Any previous systemic chemotherapy treatment, extensive brain radiotherapy, targeted therapy for locally advanced unresectable or metastatic melanoma; Immunotherapy treatment is allowed but must have ended at least 6 weeks prior to randomization.
* History of Gilbert's syndrome.
* Previous treatment with a BRAF or MEK inhibitor in metastatic setting. This treatment will be allowed in the adjuvant setting (see above). Previous treatments with immunotherapy will be allowed in both the metastatic and adjuvant setting.
* Known positive serology for human immunodeficiency virus, or an active hepatitis B or hepatitis C infection, or both.
* Impaired cardiovascular function or clinically significant cardiovascular diseases "Clinically significant (i.e., active) cardiovascular disease: cerebrovascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), a LVEF < 50% evaluated by MUGA or echocardiography, or serious cardiac arrhythmia requiring medication or a triplicate average baseline QTc interval > 500 ms."
* Uncontrolled arterial hypertension despite medical treatment.
* Moderate (Child Pugh Class B) or severe (Child Pugh Class C) hepatic impairment.
* Impairment of gastrointestinal function.
* Neuromuscular disorders associated with high concentrations of creatine kinase.
* Pregnant or nursing (lactating) women.
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study.
* Known hypersensitivity to encorafenib, binimetinib or their components.
* Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia and sensory neuropathy Grade ≤ 2 is acceptable.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 180 days after the last dose of study treatment.
* Known alcohol or drug abuse.
* Inability to swallow tablets or capsules.
* Total lactase deficiency or glucose-galactose malabsorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iván Márquez Rodaz, M.D., Study Chair — Hospital General Universitario Gregorio Marañón; Alfonso Berrocal Jaime, M.D., Study Chair — Hospital Universitario General de Valencia
Locations (21):
- Spain (21):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Institut Català d'Oncología Hospitalet, Barcelona, Barcelona, Spain
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Quirón Dexeus, Barcelona, Catalonia
  - Complejo Hospitalario Universitario Insular de Canarias, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - H. U. Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: the initial sample size was set at 48 patients, to ensure obtaining 38 evaluable patients. The cohort of symptomatic patients was exploratory and no formal sample calculation was performed, anticipating the inclusion of up to 15 patients.The trial was amended and patients were included irrespective of symptomatology.
Groups:
- COMBO450: Encorafenib - Orally, 75 mg and 50 mg capsules Binimetinib - Orally, 15 mg tablets
  In each cohort, patients will be treated with encorafenib 450 mg once daily and binimetinib 45 mg twice daily until PD or death.
  encorafenib: Encorafenib 75mg and 50mg (capsules) for a 450mg daily for oral administration during 56 days and after local radiation treatment.
  If no progression of disease progression (PD) is reported, treatment will continue until PD, unacceptable toxicity or death.
  binimetinib: Binimetinib 15mg (tablets) for a 45mg/12 hours for oral administration during 56 days and after local radiation treatment.
  Whole brain radiation therapy: The whole brain planning target volume (PTV) will receive 30 Gy in 10 fractions.
  Treatment will be delivered once daily, 5 fractions per week, over 2 to 2.5 weeks.
  Radiosurgery/stereotactic radiosurgery: Dose selection must be based on previously published Radiation Therapy Oncology Group (RTOG) data, with dose modification left up to the treating physician. The total dose will depend on the size of the metastatic lesion(s) and proximity to critical structures.
  Suggested doses are as follow: 1 fraction x 15-25 Gy; 3 fractions x 9-11 Gy; 5 fractions x 6-7 Gy; or 6 fractions x 5-6 Gy.
  For GTV > 20 mm hypofractionated stereotactic radiotherapy could be preferred. Treatment will be delivered once daily, alternate-day, 3 fractions per week.
Period: Overall Study
Arm/Group | COMBO450
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | COMBO450
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 54 [18 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 48
Eastern cooperative oncology group (ECOG) performance status (PS) at baseline [Count of Participants; unit: Participants] — The ECOG PS score describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.).
  The score ranges from 0 (Fully active, able to carry on all pre-disease performance without restriction) to 5 (dead)
  Participants
    Score 0 | 26
    Score 1 | 20
    Score 2 | 2
Barthel Index [Count of Participants; unit: Participants] — Scale used to assess a patient's functional status and monitor their progress. The scale measures a person's ability to perform 10 basic activities of daily living, thereby providing a quantitative estimate of their degree of independence. Lower values indicate worse performance and more dependency.
  Participants
    Total dependent (0-4) | 3
    Severe dependent (5-12) | 4
    Moderate dependent (13-18) | 6
    Slight dependent (19-20) | 33
    NA | 2
BRAF genotype [Count of Participants; unit: Participants] — BRAF genotype refers to changes or mutations in the BRAF gene, which is located on chromosome 7. These changes may be linked to cancer.
  Participants
    V600E: Mutated | 41
    V600E: Not mutated | 7
    V600K: Mutated | 11
    V600K: Not mutated | 37
    V600R: Mutated | 6
    V600R: Not mutated | 42
    V600 other: Mutated | 25
    V600 other: Not mutated | 23
Brain symptoms [Count of Participants; unit: Participants] — Patients who experience symptoms related to the presence of brain metastasis, including (among others):
  Headaches. Seizures. Weakness in the arms or legs. Loss of balance. Memory loss. Speech disturbance/problems talking.
  Participants
    Asymptomatic | 25
    Symptomatic | 23
Sum of longest diameters of intracranial target lesions [Median (Full Range); unit: millimeters] — This endpoint is a surrogate of the intracranial tumor burden. Here we show the sum of the longest diameter of intracranial metastasis
  millimeters | 26.5 [6 to 134]
Number of brain target lesion [Count of Participants; unit: Participants]
  1 intracranial lesion | 21
  2 intracranial lesions | 15
  3 or more intracranial lesions | 12
Extracranial metastases [Count of Participants; unit: Participants] — Presence of extracranial disease.
  Participants
    Yes | 41
    No | 7
Lactate dehydrogenase (LDH) levels [Count of Participants; unit: Participants] — LDH is determined in blood samples. this biomarker is indicative of inflammatory processes and in metastatic melanoma is considered a prognostic factor. Elevated levels of LDH are correlated with worse outcomes.
  Participants
    ≤ upper limit normal (ULN) | 26
    > ULN | 21
    Unknown | 1
Corticosteroids use at baseline [Count of Participants; unit: Participants] — Number of patients having corticosteroids at baseline. Corticcosteroids are ofter prescribed to mitigate the symptoms of brain metastasis.
  Participants
    Yes | 33
    No | 15
Corticosteroid dose [Median (Full Range); unit: milligram per day] — The corticosteroids are collected as dexametasone equivalent. Here wwe report the daily dose prescribed. Population: The dose of corticosteroids is only reported in patients receiving corticosteroids.
  milligram per day
    number analyzed (Participants) | 33
    (all) | 8 [1 to 16]
Previous anti-PD-1 based immunotherapy [Count of Participants; unit: Participants] — PD-1 inhibitors and PD-L1 inhibitors are a group of checkpoint inhibitor anticancer drugs that block the activity of PD-1 and PDL1 immune checkpoint proteins. These treatments have an anticancer effect by promoting the activation of the immune system against tumor cells.
  Participants
    Anti PD-1 | 11
    Anti PD-1 / anti CTLA-4 | 5
    No previous PD-L1 | 32
Radiotherapy received in the EBRAIN trial [Count of Participants; unit: Participants] — Type of radiation therapy scheduled during this trial. The radiotherapy type was chosen according to the principal investigator criteria and local standard procedures.
  Participants
    Radiosurgery (RS) | 10
    Fractioned stereotactic radiotherapy (FSRT) | 6
    Whole brain radiotherapy (WBRT) | 15
    None | 17

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Objective Response (iORR) by Modified RECIST 1.1 Before Local Radiotherapy Treatment in Full Dataset
Description: iORR calculated as the proportion of patient with a best overall intracranial response of complete response (CR) or partial response (PR) before local treatment according to modified RECIST 1.1.
  Modified RECIST 1.1 consists of:
  Up to 5 intracranial lesions could be selected as target lesions Target lesions might have a longest diameter ≥ 5 mm when evaluated by contrast-enhanced MRI
  This endpoint was also independently reported in patients with symptomatic and asymptomatic brain metastasis.
Time Frame: 24 months after start of treatment
Population: The endpoint is calculated for the full dataset and also in two subgroups with symptomatic or asymptomatic brain metastasis, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | COMBO450
Number analyzed (Participants) | 48
Participants
  Full analysis set: Patients with intracranial response | 34
  Full analysis set: Patients with NO intracranial response | 13
  Full analysis set: Not evaluable | 1
  Asymptomatic brain metastasis: number analyzed (Participants) | 25
  Asymptomatic brain metastasis: Patients with intracranial response | 20
  Asymptomatic brain metastasis: Patients with NO intracranial response | 5
  Asymptomatic brain metastasis: Not evaluable | 0
  Symptomatic brain metastasis: number analyzed (Participants) | 23
  Symptomatic brain metastasis: Patients with intracranial response | 14
  Symptomatic brain metastasis: Patients with NO intracranial response | 8
  Symptomatic brain metastasis: Not evaluable | 1

2. Secondary Outcome: Duration of Intracranial Response
Description: Calculated as the time from the date of first documented CR or PR to the first documented intracranial progression or death due to underlying cancer accoridng to modified RECIST 1.1, in patients with documented intracranial CR or PR before local treatment.
Time Frame: Throughout the study period, up to approximately 24 months
Population: Only patients who have an intracranial responses were analyzed for its duration.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | COMBO450
Number analyzed (Participants) | 34
months | 5.6 [3.6 to 7.5]

3. Secondary Outcome: Intracranial Progression-free Survival (iPFS) by RECIST 1.1
Description: Defined as the time from the date of inclusion to the date of the first documented intracranial disease progression or death due to any cause, whichever occurs first. PFS was determined based on tumor assessment (modified RECIST version 1.1 criteria). The local Investigator's assessments was used for analyses. Those patients who were alive and had not progressed at the last follow-up, date of progression was censored at the date of the last follow-up. Patients with no additional image test other than baseline were censored the day after inclusion.
Time Frame: Throughout the study period, up to approximately 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | COMBO450
Number analyzed (Participants) | 48
months | 8.5 [6.4 to 11.8]

4. Secondary Outcome: Extracranial Progression-free Survival (ePFS) in Both Cohorts
Description: Defined as the time from the date of inclusion to the date of the first documented extracranial disease progression or death due to any cause, whichever occurs first. PFS was determined based on tumor assessment (RECIST version 1.1 criteria). The local Investigator's assessments was used for analyses. Those patients who were alive and had not progressed at the last follow-up, date of progression was censored at the date of the last follow-up. Patients with no additional image test other than baseline were censored the day after inclusion.
Time Frame: Throughout the study period, up to approximately 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | COMBO450
Number analyzed (Participants) | 48
months | 7.7 [6.1 to 11.8]

5. Secondary Outcome: Intracranial Progression-free Rates
Description: Proportion of patients free of intracranial progression assessed by modified RECIST at 6 months (week 24), 12 months (week 48) and 24-month (week 96) considering date of inclusion estimated through Kaplan-Meier method
Time Frame: at 6 months (week 24), 12 months (week 48) and 24-month (week 96)
Measure: Number (95% Confidence Interval); unit: Percentage of patients free of PD
Arm/Group | COMBO450
Number analyzed (Participants) | 48
Percentage of patients free of PD
  6 months | 66.8 [54.4 to 82.1]
  12 months | 29.5 [18.2 to 47.6]
  24 months | 5.5 [0.9 to 32]

6. Secondary Outcome: Overall Survival
Description: Calculated as the time from date of inclusion to date of death due to any cause.
Time Frame: Throughout the study period, up to approximately 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | COMBO450
Number analyzed (Participants) | 48
months | 15.9 [10.7 to 21.4]

7. Secondary Outcome: Overall Survival Rates
Description: Proportion of of patients alive at 6 months, 12 month and 24-month considering date of inclusion estimated using Kaplan-Meier.
  Patients alive at the moment of the analysis were censored on the date of their last follow-up.
Time Frame: at 6 months, 12 month and 24-month
Measure: Number (95% Confidence Interval); unit: Percentage of patients alive
Arm/Group | COMBO450
Number analyzed (Participants) | 48
Percentage of patients alive
  6 months | 91.6 [84.1 to 99.8]
  12 months | 59.2 [46.2 to 76]
  24 months | 15.5 [6.7 to 35.8]

8. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Number of patients experiencing treatment related adverse events. These events were graded accrding to CTCAE, a scale that ranges from 0 (less intense; no event) to 5 (death) .
  Here we report the number of patients experiencing any grade toxicities and the number of patients experiencing high grade (grade 3-5) toxicities.
Time Frame: Throughout the study period, up to approximately 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | COMBO450
Number analyzed (Participants) | 48
Participants
  Any grade toxicities: Experienced Toxicity | 40
  Any grade toxicities: Do NOT experienced toxicity | 8
  Grade 3-5 toxicities: Experienced Toxicity | 12
  Grade 3-5 toxicities: Do NOT experienced toxicity | 36

9. Secondary Outcome: Change on Quality of Life at Week 8 in Both Cohorts Based on the EORTC QLQ 30 Scale
Description: The EORTC QLQ-C30 questionnaire is validated for cancer. It is composed of 30 questions or items that assess QoL. The questionnaire is structured in 5 functional scales physical functioning, daily activities, emotional functioning, cognitive functioning and social functioning), 3 symptom scales (fatigue, pain and nausea, vomiting), 1 global health status scale, and 6 independent items (dyspnea, insomnia, anorexia, constipation, diarrhea and economic impact). Values between 1 and 4 (1: not at all, 2: a little, 3: quite, 4: a lot) are assigned according to the patient's responses to the item, only in items 29 and 30 are they evaluated with a score of 1 to 7 (1: dreadful, 7: excellent).
  The scores obtained are standardized and a score between 0 and 100 is obtained, which determines the level of impact of the cancer on the patient on each of the scales. Higher values indicate better performance
Time Frame: 8 weeks
Population: Only patients who completed the quality of life questionnaires
Measure: Median (Full Range); unit: Score
Arm/Group | COMBO450
Number analyzed (Participants) | 36
Score
  Week 8 | 85.5 [48.6 to 99.4]
  Baseline | 78.4 [29.3 to 98.7]
Statistical Analysis 1: Comparison: COMBO450; Comparison between baseline and Week 8; Test type: Superiority; p = 0.015, Wilcoxon (Mann-Whitney) — pValues below 0.05 are considered statistically significant

10. Secondary Outcome: Change on Quality of Life at Week 24 in Both Cohorts Based on the EORTC QLQ 30 Scale
Description: as for outcome 9
Time Frame: 24 weeks
Population: Only patients who completed the quality of life questionnaires
Measure: Median (Full Range); unit: Score
Arm/Group | COMBO450
Number analyzed (Participants) | 26
Score
  Week 24 | 74.9 [47.3 to 97.9]
  Baseline | 78.4 [29.3 to 98.7]
Statistical Analysis 1: Comparison: COMBO450; Comparison between baseline and W24; Test type: Superiority; p = 0.754, Wilcoxon (Mann-Whitney) — pValues below 0.05 are considered statistically significant

11. Secondary Outcome: Extracranial Progression-free Rates
Description: Proportion of patients free of extracranial progression assessed by modified RECIST at 6 months (week 24), 12 months (week 48) and 24-month (week 96) considering date of inclusion estimated through Kaplan-Meier method
Time Frame: at 6 months (week 24), 12 months (week 48) and 24-month (week 96)
Measure: Number (95% Confidence Interval); unit: Percentage of patients free of PD
Arm/Group | COMBO450
Number analyzed (Participants) | 48
Percentage of patients free of PD
  6 months | 64.1 [51.4 to 79.9]
  12 months | 31.2 [19.6 to 49.6]
  24 months | 5.8 [1 to 33.8]

ADVERSE EVENTS:
Time Frame: Throughout the study period, up to approximately 24 months
Arm/Group | COMBO450
All-Cause Mortality (participants affected / at risk) | 33/48
Serious Adverse Events (participants affected / at risk) | 22/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COMBO450 (N=48)
Anaphylaxis (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 3 (3)
Pulmonary thromboembolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right pleural empyema by streptococcus constellatus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory sepsis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Amigdalitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute renal insufficiency (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Instability (Nervous system disorders) | 1 (1)
Focal seizures (Nervous system disorders) | 1 (1)
Acute pain in rib zone irradiated to legs (General disorders) | 1 (1)
Epileptic status (Nervous system disorders) | 1 (1)
Eplectic seizures (Nervous system disorders) | 1 (1)
Brain metastasis surgery (Surgical and medical procedures) | 1 (1)
Movements involuntary (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Left Hemiparesis (General disorders) | 1 (1)
Febrile syndrome of unknown origin (General disorders) | 1 (1)
Encorafenib overdose (General disorders) | 1 (1)
Digestive bleeding (Gastrointestinal disorders) | 1 (1)
Clostridium Difficile infectious diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | COMBO450 (N=48)
Nausea (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 13
Fatigue (General disorders) | 12
Fever (General disorders) | 7
Anemia (Blood and lymphatic system disorders) | 8
Alanine aminotransferase increased (Investigations) | 9
Constipation (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Aspartate aminotransferase increased (Investigations) | 8
GGT increased (Investigations) | 8
Other not specified (Skin and subcutaneous tissue disorders) | 7
Other not specified (Investigations) | 6
Asthenia (General disorders) | 5
Dysgeusia (Nervous system disorders) | 5
Other not specified (Gastrointestinal disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
CPK increased (Investigations) | 3
Other not specified (Eye disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Creatinine increased (Investigations) | 3
Lymphocyte count decreased (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03898908/Prot_SAP_000.pdf